CLINICAL TRIAL: NCT00747760
Title: The Prevalence of TSH Receptor Mutation Among the Arab Population of Israel
Brief Title: TSH Receptor Mutations Among a Consanguineous Community
Acronym: TSHR
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Dr Yardena Tenenbaum-Rakover, Director Pediatric Endocrine Unit, Ha'Emek Medical Center, Afula, Israel
Other Study IDs: 920050194; 066-2005
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2008-09-11 (Estimated); Status verified 2008-09

CONDITIONS: Hypothyroidism
Keywords: TSH Receptor, resistance TSH, Hyperthyrortropinemia
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples were taken with EDTA and Genomic DNA was extracted from peripheral mononuclear cells using the Blood Amp Kit (QIAGEN Inc., Valencia, CA)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Extended family members
- 2: Control- subjects from the same town without known thyroid diseases

SUMMARY:
Resistance to thyrotropin (RTSH) is a condition of impaired responsiveness of the thyroid gland to TSH, characterized by elevated TSH, low or normal thyroid hormone levels, and hypoplastic or normal-sized thyroid gland.

The aim of the present study was to evaluate the clinical course over time,the genotype-phenotype association and the frequency of two different TSH-receptor (TSHR) mutations in a highly consanguineous population of the town of Um-El-Fahem.

DETAILED DESCRIPTION:
Resistance to thyrotropin (RTSH) is a syndrome involving reduced sensitivity to TSH. It is characterized by elevated TSH, absence of goiter (normal or hypoplastic thyroid gland) and normal to very low levels of thyroid hormones. The TSH-receptor (TSHR) gene is located on chromosome 14q31 and it consists of extracellular, trans-membrane and intracellular domains. Mutation in the TSHR may cause either gain or loss of function of the receptor. Loss-of-function mutations are autosomal-recessively inherited and lead to a spectrum of phenotypes, ranging from mild euthyroid hyperthyrotropinemia to severe congenital hypothyroidism (CH). Insensitivity to TSH depends on both the severity and location of the TSHR mutations. Since the first report of familial euthyroid hyperthyrotropinemia caused by a TSHR mutation, several cases of loss-of-function mutations of the TSHR have been reported however only a few reports on the outcome of patients affected with TSHR mutations. Whether the condition of euthyroid hyperthyrotropinemia leads to clinical hypothyroidism, remains stable or normalizes over time has yet to be elucidated. We recently described a unique novel TSHR-inactivating mutation located at the third extracellular loop that preferentially affected the inositol phosphate (IP) pathway in three sisters of Arab-Muslim decent that presented with euthyroid hyperthyrotropinemia. Further analysis of the extended family revealed additional members with TSHR syndrome phenotype carrying two different TSHR mutations. All the affected subjects live in the same town. The aim of the present study was to evaluate the clinical course over time, the genotype-phenotype association and the frequency of these two different TSHR mutations among the highly consanguineous population of the town of Um El Fahem.

ELIGIBILITY:
Inclusion Criteria:

* Subjects belonging to extended family of the index case

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects belonging to extended family of the index case
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2005-12; Primary Completion 2006-07 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Two specific TSHR mutations | Finished

CONTACTS AND LOCATIONS:
Overall Officials: Yardena Tenenbaum-Rakover, MD, Principal Investigator — Ha'Emelk Medical Center,Afula, Israel; Samuel Refetoff, MD, Principal Investigator — The University of Chicago, Chicago, Il, USA
Locations (2):
- Samuell Refetoff, Chicago, Illinois, United States
- Ha'Emek Medical Center, Afula, Israel

REFERENCES:
- [Background] Grasberger H, Van Sande J, Hag-Dahood Mahameed A, Tenenbaum-Rakover Y, Refetoff S. A familial thyrotropin (TSH) receptor mutation provides in vivo evidence that the inositol phosphates/Ca2+ cascade mediates TSH action on thyroid hormone synthesis. J Clin Endocrinol Metab. 2007 Jul;92(7):2816-20. doi: 10.1210/jc.2007-0366. Epub 2007 Apr 24. PMID 17456567